CLINICAL TRIAL: NCT04570449
Title: Fluoxetine to Reduce Hospitalization From COVID-19 Infection (FloR COVID-19)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study timeline is not feasible
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Erika Saunders, Hershey Medical Center Manager, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00015598
Record Dates: First submitted 2020-09-29; First posted 2020-09-30 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: covid-19; fluoxetine; cytokine; anti-inflammatory; IL-6
MeSH Terms: conditions — COVID-19 | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fluoxetine (Experimental): Participants instructed to take fluoxetine 20 mg capsule orally daily for 8 weeks in the following schedule:
  Week 1 = 1 pill (20 mg), Week 2 = 2 pills (40 mg), Weeks 3-6 = 3 pills (60 mg), Week 7 = 2 pills (40 mg), Week 8 = pill (20 mg)
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Participants instructed to take fluoxetine placebo capsule matching fluoxetine orally daily for 8 weeks in the following schedule:
  Week 1 = 1 pill, Week 2 = 2 pills, Weeks 3-6 = 3 pills, Week 7 = 2 pills, Week 8 = pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — 20 mg capsule
  Arms: Fluoxetine
Drug: Placebo — fluoxetine placebo capsule
  Arms: Placebo

SUMMARY:
The current research is a pilot study to determine the feasibility of recruiting and retaining 40 participants diagnosed with COVID-19. The purpose is to observe the early use of fluoxetine (commonly known as Prozac) to reduce the severity of the COVID-19 illness. Fluoxetine is a drug that has been approved by the U.S. Food and Drug Administration (FDA) since 1987 for various mental health disorders.

DETAILED DESCRIPTION:
Morbidity and mortality resulting from COVID-19 infections are associated with multisystem organ failure due to a rapid increase in cytokine production. Fluoxetine has been shown to reduce the mechanisms that cause the cytokine storm that leads to COVID-19 fatalities.

This is a pilot study to assess feasibility of recruiting and retaining participants diagnosed with COVID-19. The purpose of this study is to observe the early use of fluoxetine treatments on illness outcome: primary outcome is hospitalization and secondary outcomes of complications including intubation and death. Additional secondary outcomes include effects on outcomes for depression and post-traumatic stress disorder, two common illnesses which may be improved by fluoxetine.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking participant
2. 18 years of age or older
3. able to give informed consent
4. Tested positive for active SARS-CoV-2 infection and

   1. It's been less than 10 days since symptoms first appeared;
   2. Fever persists for longer than 24 hours without the use of fever reducing medications; and
   3. Experiencing other symptoms of COVID-19 as described by the CDC

Exclusion Criteria:

1. Prisoner or institutionalized patient
2. Unable to give informed consent
3. Less than 18 years of age
4. Hospitalization
5. Active bleeding requiring blood products in past week
6. Diagnosed with bipolar disorder and not on mood stabilizing medication
7. Known allergy or hypersensitivity to fluoxetine
8. Currently taking a monoamine oxidase inhibitor (MAOI)
9. Currently taking an selective serotonin reuptake inhibitor (SSRI) or selective norepinephrine reuptake inhibitor (SNRI)
10. Outpatient and currently taking hydroxychloroquine
11. Known pregnancy
12. Breastfeeding
13. Known prolonged QTc, such as congenital prolonged QTc syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of hospitalization | 8 weeks
  Measures number of subjects hospitalized for COVID-19 symptoms
Physical symptoms assessed through daily checklist | 8 weeks
  The 23-item daily symptom checklist measures the presence or absence of COVID-related symptoms (e.g. shortness of breath, fever, chills) and other possible symptoms (e.g. ear pain, vomit, seizures).

SECONDARY OUTCOMES:
Rate of intubation | 8 weeks
  Measures number of subjects intubated for COVID-19 symptoms
Rate of death | 8 weeks
  Measures number of subjects who die from COVID-19 symptoms
Depressive symptoms assessed weekly | 8 weeks
  Measured using the 9-item Patient Health Questionnaire (PHQ-9) each item rated on a scale of 0-3, where 0=no depressive symptoms and 3=depressive symptoms present nearly every day. A high score indicates severe depression.
Post traumatic stress disorder symptoms assessed weekly | 8 weeks
  Measured using the 4-item SPAN assessment rated on a scale from 0-4 where 0=not at all distressing and 4=extremely distressing. A score greater than 5 indicates the presence of PTSD.
Anxiety symptoms assessed weekly | 8 weeks
  Measured using the 7-item General Anxiety Disorder Scale (GAD-7) rated from 0-3, where 0=no anxiety symptoms and 3=anxiety symptoms present nearly ever day. A high score indicates severe anxiety.
Suicidality assessed daily | 8 weeks
  Measured using the 6-item Columbia-Suicide Severity Rating Scale (C-SSRS), a semi-structured interview on the presence or absence of suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Saunders, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center Clinical Research Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Amitai M, Taler M, Carmel M, Michaelovsky E, Eilat T, Yablonski M, Orpaz N, Chen A, Apter A, Weizman A, Fennig S. The Relationship Between Plasma Cytokine Levels and Response to Selective Serotonin Reuptake Inhibitor Treatment in Children and Adolescents with Depression and/or Anxiety Disorders. J Child Adolesc Psychopharmacol. 2016 Oct;26(8):727-732. doi: 10.1089/cap.2015.0147. Epub 2016 Jan 15. PMID 26771135
- [Background] Blatteau JE, Barre S, Pascual A, Castagna O, Abraini JH, Risso JJ, Vallee N. Protective effects of fluoxetine on decompression sickness in mice. PLoS One. 2012;7(11):e49069. doi: 10.1371/journal.pone.0049069. Epub 2012 Nov 8. PMID 23145072
- [Background] Blatteau JE, de Maistre S, Lambrechts K, Abraini J, Risso JJ, Vallee N. Fluoxetine stimulates anti-inflammatory IL-10 cytokine production and attenuates sensory deficits in a rat model of decompression sickness. J Appl Physiol (1985). 2015 Dec 15;119(12):1393-9. doi: 10.1152/japplphysiol.00602.2015. Epub 2015 Oct 22. PMID 26494447
- [Background] Branco-de-Almeida LS, Kajiya M, Cardoso CR, Silva MJ, Ohta K, Rosalen PL, Franco GC, Han X, Taubman MA, Kawai T. Selective serotonin reuptake inhibitors attenuate the antigen presentation from dendritic cells to effector T lymphocytes. FEMS Immunol Med Microbiol. 2011 Aug;62(3):283-94. doi: 10.1111/j.1574-695X.2011.00816.x. Epub 2011 Jun 16. PMID 21569123
- [Background] Cai Z, Liu J, Bian H, Cai J, Jin Q, Han J. Fluoxetine, an Antidepressant Drug, Inhibited Cigarette Smoke-Induced Pulmonary Inflammation and Apoptosis in Rats. Inflammation. 2017 Aug;40(4):1375-1381. doi: 10.1007/s10753-017-0580-y. PMID 28477248
- [Background] Dong C, Zhang JC, Yao W, Ren Q, Yang C, Ma M, Han M, Saito R, Hashimoto K. Effects of escitalopram, R-citalopram, and reboxetine on serum levels of tumor necrosis factor-alpha, interleukin-10, and depression-like behavior in mice after lipopolysaccharide administration. Pharmacol Biochem Behav. 2016 May;144:7-12. doi: 10.1016/j.pbb.2016.02.005. Epub 2016 Feb 15. PMID 26892759
- [Background] Durairaj H, Steury MD, Parameswaran N. Paroxetine differentially modulates LPS-induced TNFalpha and IL-6 production in mouse macrophages. Int Immunopharmacol. 2015 Apr;25(2):485-92. doi: 10.1016/j.intimp.2015.02.029. Epub 2015 Mar 2. PMID 25744603
- [Background] Gobin V, Van Steendam K, Denys D, Deforce D. Selective serotonin reuptake inhibitors as a novel class of immunosuppressants. Int Immunopharmacol. 2014 May;20(1):148-56. doi: 10.1016/j.intimp.2014.02.030. Epub 2014 Mar 6. PMID 24613205
- [Background] Hashioka S, Klegeris A, Monji A, Kato T, Sawada M, McGeer PL, Kanba S. Antidepressants inhibit interferon-gamma-induced microglial production of IL-6 and nitric oxide. Exp Neurol. 2007 Jul;206(1):33-42. doi: 10.1016/j.expneurol.2007.03.022. Epub 2007 Mar 30. PMID 17481608
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Li XQ, Wang HM, Yang CG, Zhang XH, Han DD, Wang HL. Fluoxetine inhibited extracellular matrix of pulmonary artery and inflammation of lungs in monocrotaline-treated rats. Acta Pharmacol Sin. 2011 Feb;32(2):217-22. doi: 10.1038/aps.2010.187. Epub 2011 Jan 10. PMID 21217769
- [Background] Liu D, Wang Z, Liu S, Wang F, Zhao S, Hao A. Anti-inflammatory effects of fluoxetine in lipopolysaccharide(LPS)-stimulated microglial cells. Neuropharmacology. 2011 Sep;61(4):592-9. doi: 10.1016/j.neuropharm.2011.04.033. Epub 2011 May 11. PMID 21575647
- [Background] Liu RP, Zou M, Wang JY, Zhu JJ, Lai JM, Zhou LL, Chen SF, Zhang X, Zhu JH. Paroxetine ameliorates lipopolysaccharide-induced microglia activation via differential regulation of MAPK signaling. J Neuroinflammation. 2014 Mar 12;11:47. doi: 10.1186/1742-2094-11-47. PMID 24618100
- [Background] Lu X, Wang J, Chen X, Jiang Y, Pan ZK. Rolipram Protects Mice from Gram-negative Bacterium Escherichia coli-induced Inflammation and Septic Shock. Sci Rep. 2020 Jan 13;10(1):175. doi: 10.1038/s41598-019-56899-6. PMID 31932743
- [Background] Roumestan C, Michel A, Bichon F, Portet K, Detoc M, Henriquet C, Jaffuel D, Mathieu M. Anti-inflammatory properties of desipramine and fluoxetine. Respir Res. 2007 May 3;8(1):35. doi: 10.1186/1465-9921-8-35. PMID 17477857
- [Background] Sherkawy MM, Abo-Youssef AM, Salama AAA, Ismaiel IE. Fluoxetine protects against OVA induced bronchial asthma and depression in rats. Eur J Pharmacol. 2018 Oct 15;837:25-32. doi: 10.1016/j.ejphar.2018.08.026. Epub 2018 Aug 23. PMID 30145150
- [Background] Taraz M, Khatami MR, Dashti-Khavidaki S, Akhonzadeh S, Noorbala AA, Ghaeli P, Taraz S. Sertraline decreases serum level of interleukin-6 (IL-6) in hemodialysis patients with depression: results of a randomized double-blind, placebo-controlled clinical trial. Int Immunopharmacol. 2013 Nov;17(3):917-23. doi: 10.1016/j.intimp.2013.09.020. Epub 2013 Oct 11. PMID 24121064
- [Background] Udina M, Hidalgo D, Navines R, Forns X, Sola R, Farre M, Capuron L, Vieta E, Martin-Santos R. Prophylactic antidepressant treatment of interferon-induced depression in chronic hepatitis C: a systematic review and meta-analysis. J Clin Psychiatry. 2014 Oct;75(10):e1113-21. doi: 10.4088/JCP.13r08800. PMID 25373120
- [Background] Vollmar P, Haghikia A, Dermietzel R, Faustmann PM. Venlafaxine exhibits an anti-inflammatory effect in an inflammatory co-culture model. Int J Neuropsychopharmacol. 2008 Feb;11(1):111-7. doi: 10.1017/S1461145707007729. Epub 2007 Apr 20. PMID 17445357
- [Background] Wang L, Wang R, Liu L, Qiao D, Baldwin DS, Hou R. Effects of SSRIs on peripheral inflammatory markers in patients with major depressive disorder: A systematic review and meta-analysis. Brain Behav Immun. 2019 Jul;79:24-38. doi: 10.1016/j.bbi.2019.02.021. Epub 2019 Feb 21. PMID 30797959
- [Background] Young KC, Bai CH, Su HC, Tsai PJ, Pu CY, Liao CS, Lin YM, Lai HW, Chong LW, Tsai YS, Tsao CW. Fluoxetine a novel anti-hepatitis C virus agent via ROS-, JNK-, and PPARbeta/gamma-dependent pathways. Antiviral Res. 2014 Oct;110:158-67. doi: 10.1016/j.antiviral.2014.08.002. Epub 2014 Aug 21. PMID 25151487